CLINICAL TRIAL: NCT01664689
Title: Intraoperative and Postoperative Outcomes of Three Ophthalmic Viscosurgical Devices During Phacoemulsification
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Iladevi Cataract and IOL Research Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: OVD12
Record Dates: First submitted 2012-08-10; First posted 2012-08-14 (Estimated); Last update posted 2012-08-14 (Estimated); Status verified 2012-08

CONDITIONS: Intraoperative Performance and Postoperative Outcomes Following Cataract Surgery

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (3):
- DiscoVisc (Active Comparator): microcoaxial phacoemulsification performed with discovisc
  Interventions: Procedure: Microcoaxial Phacoemulsification
- Healon 5 (Active Comparator): microcoaxial phacoemulsification using healon 5
  Interventions: Procedure: Microcoaxial Phacoemulsification
- Celoftal (Active Comparator): microcoaxial phacoemulsification using celoftal
  Interventions: Procedure: Microcoaxial Phacoemulsification

INTERVENTIONS:
Procedure: Microcoaxial Phacoemulsification

SUMMARY:
Ophthalmic Viscosurgical Devices (OVDs) play a crucial role during phacoemulsification, by providing endothelial protection, maintaining space, as well as facilitating surgical maneuvers, including IOL implantation. Equally important is the ease of use, good visualisation and easy removal of the OVD from the eye. Currently, 3 popularly used OVDs as a single injection sufficing for surgery are: Healon 5, DiscoVisc, and Celoftal (2% hydroxypropylmethylcellulose). Whereas, there are studies showing efficacy of each of these in clinical scenarios, there is no randomized trial comparing intraoperative performance and postoperative outcomes. The aim of this study was to compare intraoperative performance and postoperative outcomes following microcoaxial phacoemulsification when using one of the three OVDs

ELIGIBILITY:
Inclusion Criteria:

* Age related, uncomplicated senile cataracts

Exclusion Criteria:

* presence of glaucoma,
* shallow anterior chamber (ACD < 2.1mm),
* pupillary dilatation < 6mm,
* extremely dense cataracts,
* posterior polar cataract,
* subluxated cataract,
* white mature cataract,
* diabetic retinopathy,
* high myopia (defined as AL > 25mm),
* uveitis, or
* previous ocular trauma/surgery.

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2011-10; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Corneal clarity on postoperative day 1 | postoperative day 1

SECONDARY OUTCOMES:
Central corneal thickness on postoperative day 1 and week 1 | day 1 and week 1

CONTACTS AND LOCATIONS:
Locations (1):
- Iladevi Cataract & IOL Research Centre, Ahmedabad, Gujarat, India